CLINICAL TRIAL: NCT00732329
Title: Effectiveness of an Optimized Home Based Occupational Therapy for Patients With Dementia.
Brief Title: Effectiveness of Home Based Occupational Therapy for Dementia.
Acronym: ERGODEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government)
Responsible Party: Principal Investigator, Dr. Matthias Schützwohl, PD Dr., Technische Universität Dresden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LT-DEMENZ-44-074
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): optimized home based occupational therapy including:
  * diagnostic assessment
  * patient-centered definition of targets involving the care giver
  * occupational therapy
  Interventions: Behavioral: Occupational Therapy
- B (No Intervention): treatment according to guidelines of German Society for Psychiatry, Psychotherapy and Nervous Diseases (DGPPN) and German Society of Neurology (DGN) without optimized occupational therapy

INTERVENTIONS:
Behavioral: Occupational Therapy — optimized home Based Occupational Therapy including:
  * diagnostic assessment
  * patient-centered definition of targets involving the care giver
  * occupational therapy
  Arms: A

SUMMARY:
The purpose of this study is to determine if a home based occupational therapy is effective in the treatment of dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Dementia (according to DSM-IV TR)
2. A score 26 to 12 on the MMSE
3. Must be 55 or older
4. Patient is living at home or therapeutical flat sharing
5. Primary care giver at least 2 days / week available at home
6. Written informed consent from patient and care giver
7. German as dominant language

Exclusion Criteria:

1. Other dementia (p.e. frontotemporal dementia, dementia with Lewy Bodies, Creutzfeldt-Jakob disease, Parkinson's disease or atypical Parkinson's syndromes
2. Dementia with relevant displaying behavioural problems (neuropsychiatric Inventory; NPI, Subscore ≥ 8)
3. Depressive episodes (Geriatric Depression Scale, GDS (short version) ≥ 6)
4. Mental disability
5. Home Based Occupational Therapy for Dementia within the last 6 months
6. Impairment of visual and/or acoustic cognition which does not allow Occupational Therapy
7. Apoplexy with movement disorders which does not allow Occupational Therapy
8. Severe physical/systemic illnesses (cardio-pulmonal, Hematological or metabolic) which do not allow participating
9. Recent history of addictive disorder
10. Intermittent intake of depressant medication, that likely causes an impairment of cognitive performance during the trial
11. Participation in another clinical trial

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Cooperative Study/Activities of Daily Living | 2 weeks, 3 and 6 months after invention or 9, 19 and 31 weeks after randomization (treatment-as-usual-group)

SECONDARY OUTCOMES:
- for patients: cognitive performance, displaying behavioural problems, satisfaction with occupational therapy, costs of occupational therapy - for family care givers: burden, medical condition, life-satisfaction | 2 weeks, 3 and 6 months after invention or 9, 19 and 31 weeks after randomization (treatment-as-usual-group)

CONTACTS AND LOCATIONS:
Overall Officials: Vjera Holthoff, Prof., Study Chair — Department of Psychiatry and Psychotherapy of University Hospital Dresden
Locations (3):
- Germany (3):
  - Department of Psychiatry and Psychotherapy, Dresden
  - Department of Psychiatry, Psychotherapy and Psychosomatic, Günzburg
  - Department for Psychiatry, Psychosomatic und Psychotherapy (of "Park-Krankenhaus Leipzig-Südost GmbH"), Leipzig